CLINICAL TRIAL: NCT02077218
Title: Assessment of Coronary Artery Disease in Asymptomatic Survivors of Allogeneic Hematopoietic Cell Transplantation (HCT): A Pilot Feasibility Study
Brief Title: Computed Tomography and Biomarker Analysis in Diagnosing Coronary Artery Disease in Asymptomatic Patients Who Have Undergone Stem Cell Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13385; NCI-2014-00419 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13385 (Other: City of Hope Medical Center)
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Cancer Survivor; Diabetes Mellitus; Hypertension
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (CT and blood biomarkers) (Experimental): Patients undergo cardiac CT and collection of blood samples for analysis of hs-CRP via quantitative immunoturbidimetry and Lp-PLA2 via ELISA.
  Interventions: Procedure: computed tomography; Other: cytology specimen collection procedure; Other: laboratory biomarker analysis; Other: questionnaire administration

INTERVENTIONS:
Procedure: computed tomography — Undergo cardiac CT
  Other Names: tomography, computed
Other: cytology specimen collection procedure — Undergo collection of blood samples
  Other Names: cytologic sampling
Other: laboratory biomarker analysis — Correlative studies
Other: questionnaire administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies computed tomography (CT) scans and biomarker analysis in diagnosing coronary artery disease (CAD) in patients who have undergone a stem cell transplant but have no symptoms of CAD. CAD is a disease in which there is a narrowing or blockage of the coronary arteries (blood vessels that carry blood and oxygen to the heart) and patients who have undergone a stem cell transplant are at an especially high risk for CAD. A CT scan involves a series of detailed pictures of areas inside the body taken from different angles. The pictures are created by a computer linked to an x-ray machine. Studying samples of blood from patients who have undergone a stem cell transplant in the laboratory may help doctors identify and learn more about biomarkers related to CAD. Using a CT scan in combination with biomarker analysis may be a better and less-invasive way to diagnose CAD.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the feasibility of using CT-based imaging and blood biomarkers for assessment of asymptomatic coronary artery disease (CAD) in survivors of allogeneic hematopoietic stem cell transplant (HCT).

SECONDARY OBJECTIVES:

I. Determine the prevalence and severity of asymptomatic CAD, as measured by CT angiography.

II. Describe the association between patient demographics (age, sex, race/ethnicity), pre-HCT chest radiation, HCT-related exposures (total body irradiation [TBI], conditioning chemotherapy), graft-versus-host disease (GvHD) and its management and cardiovascular risk factors (CVRFs) on extent of CAD.

III. Describe the association between asymptomatic CAD and candidate blood biomarkers of vessel injury and inflammation (high-sensitivity C-reactive protein [hs-CRP], lipoprotein-associated phospholipase A2 [Lp-PLA2]).

OUTLINE:

Patients undergo cardiac CT and collection of blood samples for analysis of hs-CRP via quantitative immunoturbidimetry and Lp-PLA2 via enzyme-linked immunosorbent assay (ELISA).

ELIGIBILITY:
Inclusion Criteria:

* Alive and in complete remission at time of enrollment
* Underwent allogeneic HCT after 1995
* Time between HCT and study entry: >= 2 years
* Have at least one CVRF (hypertension, diabetes, dyslipidemia) at the time of eligibility determination

Exclusion Criteria:

* History of ischemic heart disease, stroke, or cardiomyopathy/congestive heart failure
* Abnormal renal function (glomerular filtration rate [GFR] < 60 mL/min/1.73m2)
* Pregnancy
* Known allergy to intravenous (IV) contrast
* Sustained or symptomatic ventricular dysrhythmias uncontrolled with drug therapy or implantable device; significant conduction defects (i.e.: second or third degree atrioventricular block or sick sinus syndrome)
* Current clinical evidence of moderate-to-severe obstructive pulmonary disease or reactive airway diseases (i.e.: asthma) requiring therapy
* History of drug sensitivity or allergic reaction to beta-blockers
* Currently taking calcium channel blockers such as verapramil and diltiazem
* History of unrepaired severe aortic stenosis

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Feasibility, defined by the percentage of patients that enroll onto the study, successful completion of all study measurements, ability of studies to be interpreted, and achievement of the recruitment goal | Up to 9 weeks
  The current protocol will be considered feasible if: 1) >= 30% of eligible patients that are approached for participation enroll onto the study, 2) >= 75% enrolled participants successfully complete all study measurements (history/physical examination, blood draw, completion of study questionnaires, CT-imaging), 3) >= 90% of CT-based studies can be interpreted and 4) =< 100 individuals are approached to achieve recruitment goal of 20 participants.

OTHER OUTCOMES:
Prevalence of asymptomatic CAD, as measured by CT angiography | Up to 9 weeks
  Asymptomatic CAD will be defined as having either an abnormal coronary artery calcium (CAC) (>= 100 Au) or more than minimal coronary luminal stenosis (>= 30%) in any of the arteries. Descriptive statistics will be generated to characterize the extent of luminal stenosis in the study populations.
Severity of asymptomatic CAD, as measured by CT angiography | Up to 9 weeks
  Asymptomatic CAD will be defined as having either an abnormal coronary artery calcium (CAC) (>= 100 Au) or more than minimal coronary luminal stenosis (>= 30%) in any of the arteries. Descriptive statistics will be generated to characterize the extent of luminal stenosis in the study populations.
Patient demographics (age, sex, race/ethnicity) | Up to 9 weeks
  Will be evaluated using descriptive statistics.
Pre-HCT chest radiation | Up to 9 weeks
  Will be evaluated using descriptive statistics.
HCT-related exposures (TBI, conditioning chemotherapy) | Up to 9 weeks
  Will be evaluated using descriptive statistics.
Management of GvHD | Up to 9 weeks
  Will be evaluated using descriptive statistics.
CVRF-specific characteristics | Up to 9 weeks
  Will be evaluated using descriptive statistics.
Expression of hs-CRP | Up to 9 weeks
  Standard descriptive statistics will be utilized to derive the median, mean, standard deviation, and range of individual blood biomarkers in survivors with and without CAD.
Expression of Lp-PLA2 | Up to 9 weeks
  Standard descriptive statistics will be utilized to derive the median, mean, standard deviation, and range of individual blood biomarkers in survivors with and without CAD.

CONTACTS AND LOCATIONS:
Overall Officials: Saro Armenian, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States